CLINICAL TRIAL: NCT05352191
Title: Beclomethasone in Healthy Athletes, Detection in Blood and Urine, and the Effect on Aerobic Performance
Brief Title: Beclomethasone in Healthy Athletes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western Norway University of Applied Sciences (Other)
Collaborators: The Norwegian School of Sport Sciences (Unknown); The Norwegian Doping Control Laboratory (Unknown)
Responsible Party: Principal Investigator, Amund Riiser, Associate professor, Western Norway University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 123
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Performance, Detection; Doping
MeSH Terms: interventions — Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Beclomethasone (Active Comparator): 800 ug inhaled once aday for 8 days
  Interventions: Drug: Beclomethasone
- Placebo (Placebo Comparator): one pill once aday for 8 days
  Interventions: Drug: Beclomethasone

INTERVENTIONS:
Drug: Beclomethasone — inhaled 800ug

SUMMARY:
The present study aims to assess her urine concentration of beclomethasone during and after one week of use according to the World Antidoping agency's regulations. The study will assess utility of dried blood spots to detect use of beclomethasone and the effect approved use of beclomethasone has on endurance performance in healthy (non-asthmatic ) athletes.

DETAILED DESCRIPTION:
The study is a double-blinded, randomized, controlled parallel trial with participants visiting the laboratory on four separate occasions. The purpose of the first visit is to familiarize the participant with the exercise performance protocol as well as to assess a steady state oxygen consumption (VO2) at several submaximal work rates followed by a maximal VO2 (VO2max) test. For a given participant, trials on day two, three, and four will be identical conducted on the same time of day and separated by approximately one week. Beclomethasone or placebo will be delivered daily for one week from test three to test four. Urine and blood samples will be collected after testing on experimental test two and three and self-collected daily during the seven consecutive days of self-administration, and 3, 7 and 14 days after the participants stops taking medication.

Inhaled beclomethasone is approved by the World Anti-Doping Agency (WADA) for use by athletes in and out of competition. The dose used in our study is the highest single dose recommended by the Norwegian medical agency and half of the maximal daily dose recommended. Participants will inhale 800 μg beclometason or placebo using a standard inhaler (Easyhaler) used for asthma treatment. The inhaler delivers 200 μg of beclometasone with each actuation (i.e., 4 puffs/actuations gives 800 μg) with inhalation time being approximately ~1 min (12 breaths) and the manufacturer's user instructions will be followed.

The primary objective is endurance performance measured using a 20 km simulated time trial on a stationary bike. Performance will be measured time to task completion/mean power (watts) and b). Secondary objectives are the physiological response to exercise including: a) heart rate (bpm), b) minute ventilation (Lˑmin-1), c) oxygen uptake (Lˑmin-1), d) oxygen saturation (%), e) respiratory exchange ratio (RER), f) blood lactate and glucose concentration (mmolˑL-1), and f) lung function by spirometry (forced expiratory volume in 1 second, FEV1).

The first 30 participants eligible to the study will be recruited. They must be well trained cyclists and triathletes (VO2max in mLˑkg-1ˑmin-1 ≥60♂/≥50♀) aged between 18 and 35 years. Exclusion criteria include a doctor diagnosed asthma and/or the use of anti-asthmatic medications or glucocorticoids the last 12 months prior to participation. The participants must be free from chest infection for at least 4 weeks prior to assessment; and are not to be taking any medication and have no other health or medical contradictions to them taking part in the study as confirm by information provided on a physical activity readiness questionnaire.

ELIGIBILITY:
Inclusion Criteria:

Healthy Maximal oxygen uptake >60 in male and >50 in female Signed informed consent.

-

Exclusion Criteria:

Intention to compete within 3 days after last dose of medicament Asthma diagnosis Use of anti-asthmatic medication last 12 months Upper chest infection last 4 weeks Contraindication to maximal exercise Contraindication to glucocorticoids Pregnancy or possible pregnancy Failure to obtain written informed consent

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
20km cycling timetrial performance | 3 weeks
  ergometer

SECONDARY OUTCOMES:
Detection of beclometasone in urine and dried blood spots | 3 weeks
  blood and urine samples

CONTACTS AND LOCATIONS:
Overall Officials: Amund Riiser, PhD, Principal Investigator — Western Norway University of Applied Sciences

IPD SHARING:
Plan to Share IPD: No